CLINICAL TRIAL: NCT01756781
Title: A Phase 1 Randomized, Open-Label, 2-Sequence, 2-Period Crossover Study Of The Effect Of Multiple Doses Of PD-0332991 On Midazolam Pharmacokinetics In Healthy Women of Non-Childbearing Potential
Brief Title: A Drug-Drug Interaction Study To Investigate The Potential For Multiple Doses Of Palbociclib (PD-0332991) To Alter The Pharmacokinetics Of Oral Midazolam In Adult Healthy Women of Non-Childbearing Potential.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A5481012
Record Dates: First submitted 2012-12-20; First posted 2012-12-27 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
Keywords: PD-0332991; Midazolam; Drug-Drug Interaction Study; Healthy Adult Volunteer
MeSH Terms: interventions — Midazolam; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence 1 (Experimental): Subjects randomized to Sequence 1 will receive Treatment A followed by Treatment B. Treatment A is a single 2 mg oral dose of midazolam alone. Treatment B is made up of 8 daily 125 mg oral doses of PD-0332991 and a single 2 mg oral midazolam dose on day 7 immediately after the day 7 PD-0332991 dose.
  Interventions: Drug: Midazolam; Drug: PD-0332991
- Sequence 2 (Experimental): Subjects randomized to Sequence 2 will receive Treatment B followed by Treatment A with a washout of no less than 14 days in between.Treatment B is made up of 8 daily 125 mg oral doses of PD-0332991 and a single 2 mg oral midazolam dose on day 7 immediately after the day 7 PD-0332991 dose. There will be a minimum washout of 14 days prior to beginning Treatment A. Treatment A is a single 2 mg oral dose of midazolam alone.
  Interventions: Drug: Midazolam; Drug: PD-0332991

INTERVENTIONS:
Drug: Midazolam — Treatment A includes a single 2 mg oral dose of midazolam alone. Treatment B includes a single 2 mg oral midazolam dose on day 7 immediately after the day 7 PD-0332991 dose.
  Arms: Sequence 1
Drug: PD-0332991 — Treatment B includes 8 daily 125 mg oral doses of PD-0332991.
  Arms: Sequence 1
Drug: Midazolam — Treatment B includes a single 2 mg oral midazolam dose on day 7 immediately after the day 7 PD-0332991 dose.
  Treatment A includes a single 2 mg oral dose of midazolam alone.
  Arms: Sequence 2
Drug: PD-0332991 — Treatment B is made up of 8 daily 125 mg oral doses of PD-0332991.
  Arms: Sequence 2

SUMMARY:
This is a drug-drug interaction study to compare the pharmacokinetics of a 2 mg oral dose of midazolam in adult healthy women of non-childbearing potential when administered alone and when administered along with 8 daily 125 mg doses of PD-0332991. Volunteers will be randomized to one of two sequences. Volunteers in sequence 1 will receive midazolam alone in treatment period 1, followed by multiple dose PD-0332991 and midazolam in treatment period 2. Volunteers randomized to sequence 2 will receive multiple dose PD-0332991 and midazolam in treatment period 1, and following a washout period of no less than 14 days they will receive midazolam alone in treatment period 2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females of non-child bearing potential between the ages of 18 and 65 years old.
* A Body Mass Index (BMI) of 17.5 to 32.0 kg/m2 and a total body weight >50 kg (110 lbs).
* A signed informed consent document.

Exclusion Criteria:

* Any evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* A positive urine drug screen.
* Pregnant or nursing females.
* Treatment with an investigational drug within 30 days or 5 half-lives of the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Midazolam Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 0-36hrs post midazolam dose
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).

SECONDARY OUTCOMES:
Midazolam Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0-36 hrs post midazolam dose
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Maximum Observed Plasma Midazolam Concentration (Cmax) | 0-36 hrs post midazolam dose
Time to Reach Maximum Observed Plasma Midazolam Concentration (Tmax) | 0-36 hrs post midazolam dose
Plasma Decay Half-Life (t1/2) of Midazolam | 0-36 hrs post midazolam dose
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Minimum Observed Plasma Trough Concentration (Cmin) of PD-0332991 | Prior to the 6th, 7th, and 8th oral daily PD-0332991 dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, South Miami, Florida, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481012